CLINICAL TRIAL: NCT05625334
Title: A Single-dose, Open-label, Randomized, Multi-center, 2-treatment Crossover Study to Compare the Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of Acetylsalicylic Acid Powder for Oral Inhalation With Non-enteric-coated Chewable Aspirin in Healthy Adults
Brief Title: Study to Compare the Pharmacodynamics and Pharmacokinetics of Acetylsalicylic Acid Powder for Oral Inhalation With Non-enteric-coated Chewable Aspirin in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vectura, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BORA-1A-C301
Record Dates: First submitted 2022-11-01; First posted 2022-11-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: ASA; acetylsalicylic acid; cyclooxygenase-1 enzyme; oral inhalation; inhaled; myocardial Infarction
MeSH Terms: conditions — Respiratory Aspiration; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: I-ASA 100mg, then C-ASA 162mg tablet (Experimental): Treatment A: Single dose of 100 mg ASA powder for oral inhalation (I-ASA) via DPI.
  Treatment B: Single dose of 162 mg chewable non-enteric-coated Aspirin (C-ASA).
  Interventions: Drug: ASA; Drug: non-enteric-coated chewable aspirin
- Arm 2: C-ASA 162mg tablet, then I-ASA 100mg (Experimental): Treatment B: Single dose of 162 mg chewable non-enteric-coated Aspirin (C-ASA).
  Treatment A: Single dose of 100 mg ASA powder for oral inhalation (I-ASA) via DPI.
  Interventions: Drug: ASA; Drug: non-enteric-coated chewable aspirin

INTERVENTIONS:
Drug: ASA — powder for oral inhalation via a Dry Powder Inhaler (DPI)
Drug: non-enteric-coated chewable aspirin — Orally administered

SUMMARY:
The goal of this clinical trial is to compare the pharmacodynamics (PD), pharmacokinetics (PK), safety, and tolerability of acetylsalicylic acid powder for oral inhalation (i-ASA) with non-enteric-coated chewable aspirin (C-ASA) in healthy adults by demonstrating bioequivalence.

In the first treatment period, subjects will be randomized to receive either a single dose (100 mg) of I-ASA powder via a Dry Powder Inhaler (DPI) OR a single dose (162 mg) of C-ASA tablets. After a washout period, subjects will be crossed over to receive the other treatment in the second treatment period. All subjects will receive both treatments during the study. Each single dose treatment will be followed by up to 24 hours of serial post-dose PK, PD, and safety/tolerability assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 and ≤55 years of age, with BMI >18.5 and <32.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, respiratory, hematological (e.g., thrombocytopenia, neutropenia, bleeding disorders), immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Female subjects of non-childbearing potential must be:

   1. post-menopausal OR
   2. surgically sterile at least 3 months prior to dosing.
4. Sexually active female subjects of childbearing potential must be willing to use an acceptable contraceptive method throughout the study as defined in the protocol.
5. Current non-smoker: no use of tobacco or nicotine products, including any smoking cessation nicotine-containing products (i.e., nicotine replacement therapy [patch, spray, inhaler, gum, lozenge, bupropion SR, clonidine and nortriptyline], e-cigarettes, etc.) for at least 3 months prior to screening.
6. Agrees to refrain from alcohol consumption for at least 48 hours prior to admission and 48 hours after drug administration of each period.
7. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening.
2. Positive serology test results for HBsAg, HCV antibody, or HIV antigen and antibody, at screening.
3. Positive pregnancy test or lactating female subject.
4. Positive urine drug screen, urine cotinine test, or alcohol breath test.
5. Known allergic reactions, hypersensitivity or contraindications to aspirin (ASA), ibuprofen, other NSAIDs, or other related drugs, or to any excipient in the formulation.
6. Known lack of response (lack of effect) to aspirin in the past.
7. Clinically significant x-ray, ECG abnormalities or vital signs abnormalities at screening.
8. Clinically significant abnormal laboratory parameters including:

   1. Hematocrit value ≤ 32%;
   2. Platelet count <142,000 or > 450,000 platelets per µL;
   3. ALT ≥ 3 x ULN;
   4. AST ≥ 3 x ULN.
9. Subject with abnormal lung function defined by spirometric testing such that: the post bronchodilator FEV1 < 80% of predicted normal value OR FEV1/FVC ratio < 0.70.
10. Subject with current asthma defined as post-bronchodilator FEV1 > 12% increase AND > 200 ml absolute increase from pre-bronchodilator values.

Other protocol-defined I/E criteria that apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Serum thromboxane B2 (TxB2) serum concentration - Area under the effect curve (AUEC) of the % Change from baseline (CFB) in serum TxB2 concentration (TxB2 suppression) | 24 hours post-dose

SECONDARY OUTCOMES:
Proportion of subjects achieving significant inhibition of platelet aggregation (<550 Aspirin Reaction Units [ARU]) | 2 minutes post-dose
TxB2 serum concentration - AUEC of the % CFB in serum TxB2 concentration (TxB2 suppression) | 20 minutes post-dose.
TxB2 serum concentration - AUEC of the % CFB in serum TxB2 concentration (TxB2 suppression) | 30 minutes post-dose
Time to significant inhibition of platelet aggregation (<550 ARU). | assessed up to 24 hours post-dose
Peak plasma concentrations (Cmax) of ASA | pre-dose. minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 360, 480, 720 and 1440
  PK endpoints
Peak plasma concentrations (Cmax) of SA | pre-dose. minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 360, 480, 720 and 1440
  PK endpoints
Area under the plasma concentration versus time curve (AUC0-inf) | pre-dose. minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 360, 480, 720 and 1440
  PK endpoints
Area under the plasma concentration versus time curve (AUC0-t) | pre-dose. minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 360, 480, 720 and 1440
  PK endpoints
Time to peak plasma concentrations (Tmax) of ASA | pre-dose. minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 360, 480, 720 and 1440
  PK endpoints
Time to peak plasma concentrations (Tmax) of SA | pre-dose. minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 360, 480, 720 and 1440
  PK endpoints
Incidence and frequency of Adverse Events. | screening through the 7-day to follow-up period

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sinai Hospital, Baltimore, Maryland
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurbel PA, Bliden KP, Chaudhary R, Tantry US. First In-Human Experience With Inhaled Acetylsalicylic Acid for Immediate Platelet Inhibition: Comparison With Chewed and Swallowed Acetylsalicylic Acid. Circulation. 2020 Sep 29;142(13):1305-1307. doi: 10.1161/CIRCULATIONAHA.120.047477. Epub 2020 Sep 28. No abstract available. PMID 32986482